CLINICAL TRIAL: NCT00736229
Title: Intensive Exenatide Therapy in Hyperglycemic Patients Admitted to the Coronary Intensive Care Unit
Brief Title: Intravenous Exenatide in Coronary Intensive Care Unit (ICU) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saint Luke's Health System (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-206
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Hyperglycemia; Acute Coronary Syndromes; Myocardial Infarction
Keywords: hyperglycemia; acute coronary syndromes; myocardial infarction
MeSH Terms: conditions — Hyperglycemia; Acute Coronary Syndrome; Myocardial Infarction | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exenatide (Experimental): 0.05 µg/min liquid bolus of open-label exenatide followed by a constant infusion of 0.025 µg/min for 24-48 hours
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — 0.05 µg/min bolus of open-label exenatide followed by a constant infusion of 0.025 µg/min for 24-48 hours
  Other Names: Byetta

SUMMARY:
The purpose of this study is to determine the efficacy of intravenous Exenatide therapy in hyperglycemic patients admitted to the coronary intensive care unit.

DETAILED DESCRIPTION:
Diabetic patients with acute myocardial infarction (MI) have particularly poor outcomes. Clinical practice guidelines from the American College of Cardiology/American Heart Association for the treatment of patients with acute coronary syndromes call for treatment to achieve preprandial glucose <110 mg/dL, a maximum daily target <180 mg/dL, and a post-discharge hemoglobin A1c <7%. Initiation of aggressive insulin therapy is also warranted to achieve blood glucose <150 mg/dL during days 0-3 and 80-110 mg/dL when possible thereafter. To date, no studies have been conducted assessing the efficacy of intravenous exenatide administration on achieving glucose lowering in hyperglycemic coronary ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Admission to coronary ICU
* Admission blood glucose 140-299 mg/dL
* Primary cardiovascular diagnosis by attending physician
* Under primary care of cardiology service
* Age > 18 years old
* Ventilator independent
* Able to provide informed consent

Exclusion Criteria:

* Admission blood glucose < 140 or > 300 mg/dL
* Ventilator dependent
* Unconscious sedation
* Type 1 diabetes
* Known pregnancy
* Admitted to coronary ICU for right heart cath to measure hemodynamics prior to transplant
* Post transplant procedure
* Currently enrolled in another clinical trial
* Unable to provide informed consent
* Creatinine clearance < 30 mL/min
* On insulin treatment except for monotherapy with long-acting basal insulin (e.g., insulin glargine [Lantus®] or detemir [Levemir®])
* Gastroparesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Marso, MD, Principal Investigator — Mid America Heart Institute Saint Luke's Health System
Locations (1):
- Mid America Heart Institute Saint Luke's Health System, Kansas City, Missouri, United States

REFERENCES:
- [Result] Abuannadi M, Kosiborod M, Riggs L, House JA, Hamburg MS, Kennedy KF, Marso SP. Management of hyperglycemia with the administration of intravenous exenatide to patients in the cardiac intensive care unit. Endocr Pract. 2013 Jan-Feb;19(1):81-90. doi: 10.4158/EP12196.OR. PMID 23186969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment start: October 2008 Enrollment complete: June 2010 Recruitment location: Coronary Intensive Care Unit at Saint Luke's Hospital of Kansas City All eligible patients providing informed consent were assigned to a single group: exenatide infusion
Pre-assignment Details: All glucose lowering medications were discontinued prior to infusion of exenatide to study the relation between exenatide and blood glucose.
Groups:
- Exenatide: Patients were treated with a 0.05 μg/min bolus of intravenous exenatide for 30 minutes,followed by a fixed dose infusion (0.025 μg/min) for a maximum duration of 48 hours. Blood glucose values were measured hourly following commencement of infusion.
- Moderate: In September 2009, the intensive glucose control protocol in ACS patients was modified to reflect emerging data on glucose management in the ICU. From this point forward, patients with an admission blood glucose >180 mg/dL received intravenous insulin infusion to achieve a target blood glucose 100-140 mg/dL.
- Intensive: In 2008, the Mid America Heart and Vascular Institute implemented an intensive glucose control protocol using IV insulin in critically ill hyperglycemic patients hospitalized with ACS. All patients admitted with blood glucose ≥140 mg/dL received intravenous insulin infusion to achieve a target blood glucose 90-120 mg/dL. The efficacy of this protocol has been studied compared to ACS patients with admission blood glucose >140 mg/dL admitted prior to protocol implementation.
Period: Overall Study
Arm/Group | Exenatide | Moderate | Intensive
Started | 40 (Actively Enrolled) | 71 (Historic control) | 84 (Historic Control)
Completed | 40 (All patients received bolus and fixed infusion of study drug, thus completed the study) | 71 | 84
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide | Moderate | Intensive | Total
Number analyzed (Participants) | 40 | 71 | 84 | 195
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 41 | 45 | 107
  >=65 years | 19 | 30 | 39 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11.9) | 64 (11.5) | 64 (13.7) | 64.18 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 26 | 32 | 65
  Male | 33 | 45 | 52 | 130
Region of Enrollment [Number; unit: participants]
  United States | 40 | 71 | 84 | 195

OUTCOME MEASURES:

1. Primary Outcome: Median Glucose Values From Steady State Through 48 Hours or Until Discharge.
Description: Time to steady state was defined as the time from the initiation of drug infusion to first glucose value that is ≤140 mg/dl. Median glucose values were then calculated for each patient from the start of steady state through 48 hours or until discharge.
Time Frame: 1-48 hours
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: mg/dL
Groups:
- Exenatide: Patients with admission blood glucose values of 140-400 mg/dL admitted to the coronary intensive care unit were eligible. Patients that provided consent were intravenously infused with Exenatide as a 0.05 mcg/min bolus for 30 minutes followed by a fixed 0.025 mcg/min dose for up to 48 hours. Blood glucose values were measured hourly following commencement of infusion.
- Moderate: In September 2009, the intensive glucose control protocol in acute coronary syndrome (ACS) patients was modified to reflect emerging data on glucose management in the ICU. From this point forward, all patients with an admission blood glucose >180 mg/dL received intravenous insulin infusion to achieve a target blood glucose 100-140 mg/dL. These data came from a medical record review and the retrospective data collection and analysis were approved by the Saint Luke's Hospital Institutional Review Board.
- Intensive: In 2008, the Mid America Heart and Vascular Institute implemented an intensive glucose control protocol using IV insulin in critically ill hyperglycemic patients hospitalized with ACS. All patients admitted with blood glucose ≥140 mg/dL received intravenous insulin infusion to achieve a target blood glucose 90-120 mg/dL. The efficacy of this protocol has been studied compared to ACS patients with admission blood glucose >140 mg/dL admitted prior to protocol implementation. These data came from a medical record review and the retrospective data collection and analysis were approved by the Saint Luke's Hospital Institutional Review Board.
Arm/Group | Exenatide | Moderate | Intensive
Number analyzed (Participants) | 40 | 71 | 84
mg/dL | 132 [110 to 157] | 127 [105 to 161] | 105 [92 to 128]
Statistical Analysis 1: Comparison: Exenatide vs Moderate vs Intensive; Median Glucose Values (mg/dl) after steady state were evaluated across the three groups (Exenatide,Moderate and Intensive) with a Kruskal-Wallis test; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis — Comparison for the difference in Median glucose values during steady state across all three groups
Statistical Analysis 2: Comparison: Exenatide vs Intensive; Median Glucose Values (mg/dl) after steady state were evaluated between the Exenatide and Intensive study groups using a Wilcoxon Rank Sum tests; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — Comparison of Median Glucose Values between Exenatide and Intensive Groups
Statistical Analysis 3: Comparison: Exenatide vs Moderate; Median Glucose Values (mg/dl) after steady state were evaluated between the Exenatide and Moderate study groups using a Wilcoxon Rank Sum tests; Test type: Superiority or Other; p = 0.15, Wilcoxon (Mann-Whitney) — Comparison of Median Glucose Values between Exenatide and Moderate Groups

2. Primary Outcome: Time to Steady State
Description: Time to steady state was defined as the time from the initiation of drug infusion (Exenatide or Insulin) to first glucose value that is ≤140 mg/dl.
Time Frame: Start of infusion through 48 hours or until discharge
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Exenatide | Moderate | Intensive
Number analyzed (Participants) | 40 | 71 | 84
hours | 2.0 [1.5 to 5.0] | 12.0 [7.0 to 15.0] | 3.0 [1.0 to 5.0]
Statistical Analysis 1: Comparison: Exenatide vs Moderate vs Intensive; Median Time (Hrs) to steady state was evaluated across the three groups (exenatide, moderate and intensive) with a Kruskal-Wallis test; Test type: Superiority or Other; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Exenatide vs Intensive; Median time (hours) to steady state were evaluated between the Exenatide and Intensive study groups using a Wilcoxon Rank Sum tests; Test type: Superiority or Other; p = 0.80, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Exenatide vs Moderate; Median time (hours) to steady state were evaluated between the Exenatide and Moderate study groups using a Wilcoxon Rank Sum tests; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Rates of Hypoglycemia and Severe Hypoglycemia
Description: Total number of patients having at least one hypoglycemic episode (blood glucose less than 70 mg/dl), including episodes classified as severe (blood glucose less than 50 mg/dl)
Time Frame: 1-48 hours
Measure: Number; unit: participants
Arm/Group | Exenatide | Moderate | Intensive
Number analyzed (Participants) | 40 | 71 | 84
participants
  Patients with at least one hypoglycemic episode | 4 | 14 | 22
  Patients with at least one severe episode | 0 | 2 | 1

4. Secondary Outcome: Serious Adverse Events (Death, Non-fatal Myocardial Infarction, and Non-fatal Stroke Through 30 Days)
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Exenatide
Number analyzed (Participants) | 40
participants | 4

ADVERSE EVENTS:
Time Frame: Until hospital discharge or a maximum of 48 hrs, whichever was shorter.
Description: Patients were continually monitored from study drug start until discharge to collect serious and other adverse events.
Arm/Group | Exenatide
Serious Adverse Events (participants affected / at risk) | 4/40
Other Adverse Events (participants affected / at risk) | 6/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=40)
Death (Cardiac disorders) | 3 (3)
Stroke (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=40)
Vomiting (Gastrointestinal disorders) | 2 (2)
Drug failure (Metabolism and nutrition disorders) | 3 (3) — If at anytime after 6 hours of study drug administration there are four consecutive fingerstick glucose levels greater than 200 mg/dL the nurse caring for participant will classify drug failure.
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Modest number of patients enrolled, not powered to examine the effects of exenatide on hard clinical outcomes, no randomization, differences in baseline glucose levels and duration of therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No